CLINICAL TRIAL: NCT02123771
Title: Gamma-Glutamyl Transpeptidase (GGT): A Potential Diagnostic Marker for Helicobacter Pylori Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Gastroenterology & Hepatology, Prof Yeoh Khay Guan, National University Hospital, Singapore
Other Study IDs: 2011/00113
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Focus of Study : HELICOBACTER PYLORI INFECTIONS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples(solid/semi-solid) between 1-5 g will be collected and tested using ELISA for the presence of the H. pylori GGT antigen using monoclonal antibodies against GGT.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Helicobactor Pylori Infection: Comparison on the presence/absence of GGT antigen in the stool will be compared between H. pylori-positive and H. pylori-negative subjects. Rapid urease test result from the respective patients will be used as the golden standard. Should the GGT antigen in stool samples show promise in distinguishing between H. pylori-infected and uninfected individuals, sensitivity and specificity of the stool antigen test can then be established.

SUMMARY:
The investigators hypothesis:

Presence of anti-GGT (antibody against GGT) indicates H. pylori infection.

DETAILED DESCRIPTION:
Subjects will be requested to provide 1-5g of their solid/semi-solid stool sample, to be collected within 24 hours prior to their scheduled visit for urea breath test. Patients should not have been treated for H. pylori prior to stool collection. Stool samples will be tested using ELISA for the presence of the H. pylori GGT antigen using monoclonal antibodies against GGT. Stool samples will also be tested for the presence of H. pylori DNA using PCR and Western blot analysis respectively.

Presence of the GGT antigen in stool will be compared between H. pylori-positive and H. pylori-negative patients. Rapid urease test results will be used as the gold standard of H. pylori diagnosis. The sensitivity and specificity of the stool antigen test will be established.

ELIGIBILITY:
Inclusion Criteria:

* The subject is greater than 21 years of age.
* The subject must have personally signed and dated the patient informed consent form indicating that he/she has been informed of all pertinent aspects of the study.
* The subject must be willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* Subjects who have been taking antibiotics over the past 1 month will be excluded from study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients seen in Gastro clinic will be recruited for this study. Patient should 21 years and above and agreeable for study. Patient should not have been treated for H. pylori prior to stool collection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Stool anti-GGT for the diagnosis of Helicobactor Pylori Infection | 1 month after stool samples collected
  1-5g of stool samples will also be collected from patients recruited to this study, in a preliminary investigation to determine the sensitivity and specificity of a stool H.pylori antigen test.
  Rapid urese test is the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Guan Lim, Principal Investigator — NUHS
Locations (1):
- Nuhs Umc/Udc, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Gong M, Ling SS, Lui SY, Yeoh KG, Ho B. Helicobacter pylori gamma-glutamyl transpeptidase is a pathogenic factor in the development of peptic ulcer disease. Gastroenterology. 2010 Aug;139(2):564-73. doi: 10.1053/j.gastro.2010.03.050. Epub 2010 Mar 27. PMID 20347814